CLINICAL TRIAL: NCT02385890
Title: Pulse EnRiched Food and Exercise Clinical Trials (PERFECT Project): Part 1 - Acute Effects of Pulse Ingredients in Snack Products on Appetite, Blood Glucose, and Food Intake in Adults - Study 3
Brief Title: PERFECT Project - Part 1 - Study 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Alberta Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2014:114-5
Record Dates: First submitted 2014-12-17; First posted 2015-03-11 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Prevention; Obesity Prevention
MeSH Terms: interventions — Pea Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Bagel control (Experimental): 100% wheat flour
  Interventions: Other: Control
- Bagel with pea flour (Experimental): Pea flour
  Interventions: Other: Pea flour
- Bagel with pea fibre (Experimental): Pea fibre
  Interventions: Other: Pea fibre
- Bagel with pea protein (Experimental): Pea protein
  Interventions: Other: Pea protein
- Bagel with pea flour + pea protein (Experimental): Pea flour + pea protein
  Interventions: Other: Pea flour + pea protein
- Bagel with pea fibre + pea protein (Experimental): Pea fibre + pea protein
  Interventions: Other: Pea fibre + pea protein

INTERVENTIONS:
Other: Control — Non pulse ingredient bagel
  Arms: Bagel control
Other: Pea flour — Pulse ingredient bagel
  Arms: Bagel with pea flour
Other: Pea fibre — Pulse ingredient bagel
  Arms: Bagel with pea fibre
Other: Pea protein — Pulse ingredient bagel
  Arms: Bagel with pea protein
Other: Pea flour + pea protein — Pulse ingredient bagel
  Arms: Bagel with pea flour + pea protein
Other: Pea fibre + pea protein — Pulse ingredient bagel
  Arms: Bagel with pea fibre + pea protein

SUMMARY:
The objectives are to test the acute effects of different bagels containing pulse ingredients on: 1) post-prandial blood glucose, insulin and appetite for two hours, and 2) food intake two hours following consumption of pulse products.

The investigators hypothesize that bagels containing pulse ingredients will lead to lower blood glucose, insulin, appetite and food intake responses compared to non-pulse bagels.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L) and normotensive (systolic blood pressure <140 mm Hg and diastolic blood pressure below < 90 mm Hg)
* BMI of 18.5-29.9 kg/m2

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Those who are active (organized activities or athletic training at a high intensity; ≥ 150 min per week of moderate to vigorous physical activity)
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year.
* Those unable to walk for an hour continuously

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose and Insulin Concentrations | 0-200
  Measured in blood using intravenous catheter at 12 time points used to calculate area under curve (AUC). Glucose will be determined by automated methods using Abbot Spectrum CCX Analyzer, and Insulin will be measured by commercially available RIA kits
Food Intake | at 120 min
  Ad-libitum meal. Food consumed measured by weight
Subjective Appetite | 0-200 min
  Motivation-to-eat VAS questionnaire used to calculate area under curve (AUC)

SECONDARY OUTCOMES:
Palatability of meal | at 140 mins
  Measured by VAS questionnaire
Palatability of treatments | at 5 mins
  Measured by VAS questionnaire
Physical comfort | 0 - 200 min
  Measured by VAS questionnaire at 12 time points used to calculate area under curve (AUC)
Energy/fatigue measured by VAS questionnaire | 0 - 200 mins
  Measured by VAS questionnaire at 12 time points, used to calculate area under curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada